CLINICAL TRIAL: NCT03210285
Title: Whole Exome Sequencing (WES) of NF2-associated in Comparison to Sporadic Vestibular Schwannomas - Correlation With Clinical Data
Brief Title: WES of NF2-associated in Comparison to Sporadic Vestibular Schwannomas - Correlation With Clinical Data
Acronym: NF2
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Sponsor
Other Study IDs: NF2Tue
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2017-07

CONDITIONS: Neurofibromatosis Type 2; Vestibular Schwannoma; Acoustic Neuroma
Keywords: Whole exome sequencing; Neurofibromatosis Type 2; Acoustic Neuroma; Vestibular schwannoma
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic | interventions — Exome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tumor tissue Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NF2-associated VS: Patients after surgery of a NF2- associated vestibularis schwannoma: Whole exome sequencing of blood and tumor tissue
  Interventions: Diagnostic Test: Whole exome sequencing
- Sporadic VS: Patients after surgery of a sporadic vestibularis schwannoma: : Whole exome sequencing of blood and tumor tissue
  Interventions: Diagnostic Test: Whole exome sequencing

INTERVENTIONS:
Diagnostic Test: Whole exome sequencing — Whole exome sequencing

SUMMARY:
Whole exome sequencing (WES) of 50 sporadic and 50 Neurofibromatosis Type2 (NF2)-associated vestibularis schwannomas (VS) in children and young adults. The aim is to gain insight into the complete genome of the NF2 associated VS compared to sporadic VS (control group). These data are to be correlated with the clinic, ie the auditory function (audiogram, acoustically evoked potentials) and the clinical picture as well as the tumor growth rate and general data such as sex, age, side, etc.

DETAILED DESCRIPTION:
Whole exome sequencing (WES) of 50 sporadic and 50 Neurofibromatosis Type2 (NF2)-associated vestibularis schwannomas (VS) in children and young adults. The aim is to gain insight into the complete genome of the NF2 associated VS compared to sporadic VS (control group). These data are to be correlated with the clinic, ie the auditory function (audiogram, acoustically evoked potentials) and the clinical picture as well as the tumor growth rate and general data such as sex, age, side, etc.

The analysis of genetic changes should provide a better insight into the oncogenesis of these tumors. The distinct genetic characteristics between NF2-associated and sporadic VS suggest a different oncogenesis of these tumors.

The correlation of the genetic characteristics with the partly very different clinical appearance and a very different dynamics of the disease, in particular the tumor volume in the course, identifies the underlying modifiers of the disease course.

Based on these genetic modifiers, patients can be stratified and individual clinical therapy decisions can be made.

By demonstrating these genetic profiles in the peripheral blood, prospective conclusions can be drawn about expected disease progression before intervention as well as for therapy monitoring

ELIGIBILITY:
Inclusion Criteria:

* Study population: Operated NF2-associated VS
* Control group: Operated sporadic VS
* Consent to participation in the study by the patient / legal guardian in prospective inclusion or consent to the use of stored specimens in retrospective inclusion
* Age: 0 -99 years

Exclusion Criteria:

* Lack of informed consent
* Patient's request (withdrawal of the consent statement for the evaluation of the data and further storage of the blood / tissue samples)

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Study population: Operated NF2-associated VS
  * Control group: Operated sporadic VS
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation clinical-volumetric pathologies and distinct genetic features | Within 1 week after measurement
  Correlation between interindividually different clinical-volumetric pathologies and distinct genetic features

SECONDARY OUTCOMES:
Identification of genetic profiles for pre-interventional prediction of expected disease progression | Within 1 week after measurement
  Identification of genetic profiles in the peripheral blood for pre-interventional prediction of expected disease progression as well as therapy monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuhmann, Prof. Dr., Study Director — University Hospital Tübingen
Locations (1):
- University Department of Neurosurgery Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No